CLINICAL TRIAL: NCT02555644
Title: A Phase 1b Trial of LY2606368 in Combination With Chemoradiation in Patients With Locally Advanced Head and Neck Squamous Cell Cancer
Brief Title: A Study of Prexasertib (LY2606368) With Chemotherapy and Radiation in Participants With Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16016; I4D-MC-JTJI (Other: Eli Lilly and Company); 2015-001215-12 (EudraCT Number)
Record Dates: First submitted 2015-09-18; First posted 2015-09-21 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02-01

CONDITIONS: Head and Neck Neoplasms
Keywords: cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — prexasertib; Cisplatin; Cetuximab; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prexasertib + Cisplatin + Radiation Therapy (Part A) (Experimental): Prexasertib administered intravenously (IV) every 14 days over an approximately 49-day treatment period.
  Cisplatin administered IV every 7 days over an approximately 49-day treatment period.
  Intensity modulated radiation therapy administered 5 days per week over an approximately 49-day treatment period.
  Participants may remain on treatment until completion of the treatment period.
  Interventions: Drug: Prexasertib; Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy
- Prexasertib + Cetuximab + Radiation Therapy (Part B) (Experimental): Prexasertib administered IV every 14 days over an approximately 56-day treatment period.
  Cetuximab administered IV every 7 days over an approximately 56-day treatment period.
  Intensity modulated radiation therapy administered 5 days per week over an approximately 56-day treatment period (starting at Week 2).
  Participants may remain on treatment until completion of the treatment period.
  Interventions: Drug: Prexasertib; Drug: Cetuximab; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Drug: Prexasertib — Administered IV
  Other Names: LY2606368
Drug: Cisplatin — Administered IV
  Arms: Prexasertib + Cisplatin + Radiation Therapy (Part A)
Drug: Cetuximab — Administered IV
  Other Names: Erbitux; LY2939777
  Arms: Prexasertib + Cetuximab + Radiation Therapy (Part B)
Radiation: Intensity Modulated Radiation Therapy

SUMMARY:
The main purpose of this study is to investigate the safety of prexasertib in combination with other anti-cancer drugs (cisplatin or cetuximab) and radiation therapy in participants with locally advanced head and neck cancer. The study has two parts (A and B). Participants will only enroll in one part.

DETAILED DESCRIPTION:
The primary purpose of Parts A and B of this study is to determine a recommended dose level of prexasertib (an inhibitor of checkpoint kinase 1[Chk-1]) in combination with cisplatin and radiation therapy (Part A) or cetuximab and radiation therapy (Part B) in participants with locally advanced head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to comply with the treatment plan and follow-up schedule
* Must have diagnosis of head and neck squamous cell carcinoma of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal walls), hypopharynx, or larynx
* Have adequate organ function
* If participant is of reproductive potential, must agree to use medically approved contraceptive precautions during the study and for six months following the last dose of study drug
* If the participant is a female of childbearing potential, must have had a negative serum or urine pregnancy test within 14 days of the first dose of study drug and must not be breast feeding

Exclusion Criteria:

* Must not have taken an unapproved drug as treatment for any indication within the last 28 days prior to starting study treatment
* Must not have received any of the following prior therapies or treatments: systemic therapy for the study cancer, radiation therapy to the head and neck region, or curative-intent surgery in the head and neck region
* Have evidence of a distant metastatic disease
* Must not have an active symptomatic fungal, bacterial or viral infection, including human immunodeficiency virus (HIV) or Hepatitis A, B, or C
* Must not have a serious heart condition, such as congestive heart failure, unstable angina pectoris, or heart attack within the last three months
* Must not have a family history of long corrected QT interval (QTc) syndrome
* Must not have known allergic reaction against any of the components of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-02-24 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Part A: Maximum Tolerated Dose of Prexasertib in Combination with Cisplatin and Radiation Therapy | First Dose through Last Dose (Estimated up to 7 Weeks)
Part B: Maximum Tolerated Dose of Prexasertib in Combination with Cetuximab and Radiation Therapy | First Dose through Last Dose (Estimated up to 8 Weeks)

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration of Prexasertib, Cisplatin and Cetuximab | First Dose through Last Dose (Estimated up to 8 Weeks)
PK: Area Under the Concentration Curve (AUC) of Prexasertib | First Dose through Last Dose (Estimated up to 8 Weeks)
Locoregional Control Rate | Baseline through One Year (Estimated as up to 52 Weeks) or Death from Any Cause

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (2):
  - University of Alabama at Birmingham Medical Center, Birmingham, Alabama
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- France (2):
  - Centre Leon Berard, Lyon
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Zeng L, Nikolaev A, Xing C, Della Manna DL, Yang ES. CHK1/2 Inhibitor Prexasertib Suppresses NOTCH Signaling and Enhances Cytotoxicity of Cisplatin and Radiation in Head and Neck Squamous Cell Carcinoma. Mol Cancer Ther. 2020 Jun;19(6):1279-1288. doi: 10.1158/1535-7163.MCT-19-0946. Epub 2020 May 5. PMID 32371584
- [Derived] Zeng L, Beggs RR, Cooper TS, Weaver AN, Yang ES. Combining Chk1/2 Inhibition with Cetuximab and Radiation Enhances In Vitro and In Vivo Cytotoxicity in Head and Neck Squamous Cell Carcinoma. Mol Cancer Ther. 2017 Apr;16(4):591-600. doi: 10.1158/1535-7163.MCT-16-0352. Epub 2017 Jan 30. PMID 28138028
- See also: Click here for more information about this study: A Study of Prexasertib (LY2606368) with Chemotherapy and Radiation in Participants with Head and Neck Cancer — http://www.lillytrialguide.com/EN/studies/cancer/jtji